CLINICAL TRIAL: NCT04312919
Title: Cleveland Clinic Families Get Fit (CCFit) : A Family-based Activity-Monitor Intervention in Pediatric Obesity
Acronym: CCFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Andrea Mucci, Associate Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-1339
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 3 in-person visit group
  Interventions: Behavioral: Family Based Activity Intervention
- Control/Crossover Group (Active Comparator): 5 in-person visit group
  Interventions: Behavioral: Family Based Activity Intervention

INTERVENTIONS:
Behavioral: Family Based Activity Intervention — Providing youth and their families with access to the knowledge and resources to increase their physical activity will allow them to lead more healthy lifestyles will provide them with the foundation for a healthier life, and future ahead.

SUMMARY:
This is a randomized prospective study to evaluate the effectiveness of a family-based intervention using activity-monitors (I.e. Fitbits) in children and adolescents aged 8-18 years with a BMI greater than or equal to 95%ile who attend the Cleveland Clinic multidisciplinary "Be Well" pediatric obesity clinic.

ELIGIBILITY:
Inclusion Criteria:

* Be Well patient
* Age 8*-18 years
* BMI > 95%ile
* English speaking

Exclusion Criteria:

* Uncontrolled asthma
* Orthopedic or other medical issue limiting mobility
* Participant has worn an activity-monitor in the past 6 months (ok if parents wear)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | Change from Baseline Six Minute Walk Distance through study completion (up to 33 weeks)
  6 minute walk distance

SECONDARY OUTCOMES:
Weight | Change from Baseline weight through study completion (up to 33 weeks)
  weight measured in kilograms
Fitbit Data | Change in steps per day wearing Fitbit and after 1 week Goal Setting Steps
  Steps per Day
Height | Change from Baseline height through study completion (up to 33 weeks)
  height measured in centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States